CLINICAL TRIAL: NCT06518356
Title: Investigating the Direct Brain Effects of Activating the Auricular Branch of the Vagus Nerve From the Cymba Concha or Mastoid Process: a Sham-controlled fMRI Study
Brief Title: Mastoid taVNS-fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Xiaolong Peng, Research Instructor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00137424
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Auricular Stimulation
Keywords: Healthy Volunteer Studies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- Auricular Neurostimulation (Active 1) (Active Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -Cymba stimulation (15Hz stimulation of cymba conchae)
  Interventions: Device: Transcutaneous Auricular Neurostimulation (tAN)
- Auricular Neurostimulation (Active 2) (Active Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -Mastoid stimulation (15Hz stimulation of mastoid process)
  Interventions: Device: Transcutaneous Auricular Neurostimulation (tAN)
- Auricular Neurostimulation (Sham 1) (Sham Comparator): •Within the MRI scanner, each participant will be connected to a series of tAN electrodes that stimulate the following ear target
  -Sham (15Hz stimulation of the earlobe)
  Interventions: Device: Transcutaneous Auricular Neurostimulation (tAN)

INTERVENTIONS:
Device: Transcutaneous Auricular Neurostimulation (tAN) — The intervention the investigators are studying is called transcutaneous auricular neurostimulation (tAN). tAN is simply electrical nerve stimulation administered at the ear which targets the auricular branch of the vagus nerve (ABVN) at the cymba conchae and mastoid process, and to a sham site (earlobe).

SUMMARY:
The purpose of this study is to explore whether stimulating different outer parts of the ear using a non-invasive form of ear stimulation called transcutaneous auricular vagus nerve stimulation (taVNS) will create different brain activation images. Investigators will recruit 24 healthy participants. The ear stimulation will be delivered while taking brain images using a magnetic resonance imaging (MRI) machine.

DETAILED DESCRIPTION:
Transcutaneous auricular vagus nerve stimulation (taVNS) is a non-invasive neuromodulation technique that delivers electric stimulation to the auricular branch of the vagus nerve (ABVN). This technique has been demonstrated effective in the treatment of depression and addiction in previous studies.

Most previous applications of taVNS targeted the ABVN via the cymba conchae or tragus sites. The mastoid process (mastoid site) is an important dermatome innervated by the ABVN, but there is currently a lack of knowledge on how taVNS on the mastoid site affects brain activity and whether it differs from the effect of stimulating the cymba site.

In this proposed study, the investigators plan to explore whether delivering taVNS to the mastoid site and the cymba site can induce different patterns of brain activity. Ultimately, if successful, this project will not only deepen our knowledge in basic neuroscience but also have great value in clinical applications since the mastoid site is a much more accessible ABVN target compared to other sites.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have the capacity and ability to provide one's own consent in English and sign the informed consent document.

Exclusion Criteria:

* Unable to speak in English.
* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions
* Metal implant devices in the head, heart or neck.
* History of brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Participant has abnormal ear anatomy, skin irritation, or ear infection present
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of psychosis or mania, or individuals who are actively manic or psychotic.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level-dependent (BOLD) signal changes during stimulation relative to sham stimulation | 30 minutes
  taVNS will be administered to participants within the bore of the MRI scanner while the investigators acquire high-resolution functional neuroimaging. Both a general linear model and SNM approach will be used to examine BOLD signal changes during stimulation relative to rest blocks, comparing each of the 3 stimulation targets within- and between- subjects to identify any differences in brain activity during stimulation of the mastoid site compared to the cymba site and sham site.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Peng, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No